CLINICAL TRIAL: NCT00400660
Title: First Time in Human, Single Dose and Repeat Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of GSK615915
Brief Title: A First Time In Human Study To Assess The Compound GSK615915
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: OLA103920
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Bronchospasm
Keywords: GSK615915 asthma surfactant MDI
MeSH Terms: conditions — Bronchial Spasm

ARMS (6):
- Subjects receiving treatment sequence 1: Part 1 (Experimental): Eligible subjects will receive placebo followed by GSK615915A with a starting dose of 250 micrograms.
  Interventions: Drug: GSK615915A; Drug: Placebo
- Subjects receiving treatment sequence 2: Part 1 (Experimental): Eligible subjects will receive GSK615915A with a starting dose of 250 micrograms followed by placebo.
  Interventions: Drug: GSK615915A; Drug: Placebo
- Subjects receiving treatment sequence 1: Part 2 (Experimental): Eligible subjects will receive placebo followed by GSK615915A with a starting dose of 250 micrograms.
  Interventions: Drug: GSK615915A; Drug: Placebo
- Subjects receiving treatment sequence 2: Part 2 (Experimental): Eligible subjects will receive GSK615915A with a starting dose of 250 micrograms followed by placebo.
  Interventions: Drug: GSK615915A; Drug: Placebo
- Subjects receiving GSK615915A: Part 3 (Experimental): Eligible subjects will receive GSK615915A with a starting dose of 250 micrograms.
  Interventions: Drug: GSK615915A
- Subjects receiving placebo: Part 3 (Experimental): Eligible subjects will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK615915A — GSK615915A inhaler will be given with a dose of 250 micrograms per metered actuation and 120 actuations per inhaler.
  Arms: Subjects receiving GSK615915A: Part 3; Subjects receiving treatment sequence 1: Part 1; Subjects receiving treatment sequence 1: Part 2; Subjects receiving treatment sequence 2: Part 1; Subjects receiving treatment sequence 2: Part 2
Drug: Placebo — Subjects will also receive placebo inhaler.
  Arms: Subjects receiving placebo: Part 3; Subjects receiving treatment sequence 1: Part 1; Subjects receiving treatment sequence 1: Part 2; Subjects receiving treatment sequence 2: Part 1; Subjects receiving treatment sequence 2: Part 2

SUMMARY:
GSK615915A is being developed as a novel surfactant for use in the formulation of GSK's future generation of Metered Dose Inhalers (MDIs). A surfactant in a MDI would provide a more stable drug suspension, this in turn will produce a consistent dose of drug being delivered with each puff.

ELIGIBILITY:
Inclusion Criteria:

* Women of non-child bearing potential.
* Body weight = 50 kg (110 lbs) for men and = 45 kg for women and Body Mass Index (BMI) within the range 19.0-30.0 kg/m²
* The subject is a current non-smoker who has not used any tobacco products in the last 12 months with a pack history of = 10 pack years.
* The subject has demonstrated the ability to correctly use a metered dose inhaler device.
* If asthmatic:

The subject must be clinically stable The subject has a baseline FEV1 = 80% of predicted.

Exclusion Criteria:

* As a result of the medical interview, physical examination or screening investigations, the Physician Responsible considers the volunteer unfit for the study.
* The subject has a history of allergy to excipients, MDI propellants, or a history of drug or other allergy that, in the opinion of the physician responsible makes the volunteer unfit to participate.
* The subject has recently participated in another clinical trial.
* The subject has used prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St Johnâ€™s Wort) within 7 or 14 days.
* The subject has an average weekly alcohol intake of greater than 21 units if male or 14 units if female, or an average daily intake of greater than 3 units regularly, where 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* Any history of breathing problems (e.g. history of asthmatic symptoms).
* The subject is infected with the hepatitis B, hepatitis C, or HIV virus.
* The subject is has a positive drugs of abuse test.
* The subject has had a respiratory tract infection within 4 weeks of the start of the study.
* The subject has a past or present disease, which as judged by the Doctor, may affect the outcome of this study.
* The subject has a history of life-threatening asthma.
* The subject has taken inhaled, nasal or dermal steroids within 4 weeks or oral steroids within 8 weeks of the start of the study.
* The subject has taken long acting inhaled beta 2 agonists within 96 hours before the screening visit.
* The subject has taken short acting inhaled beta 2 agonists within 8 hours before the screening visit.
* The subject is unable to abstain from other drugs that may interfere with the conduct of the study or its interpretation.
* The subject has ongoing rhinitis that requires treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2005-11-23 (Actual); Primary Completion 2006-07-03 (Actual); Study Completion 2006-07-03 (Actual)

PRIMARY OUTCOMES:
Side effects Lung function Blood tests Heart rate and blood pressure Heart monitored (ECG) | Up to 18 weeks

SECONDARY OUTCOMES:
Levels of GSK615915A and any breakdown products in the blood and urine. | Up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Edinburgh, West Lothian, United Kingdom

REFERENCES:
- See also: Results for study OLA103920 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/OLA103920?search=study&study_ids=OLA103920#rs